CLINICAL TRIAL: NCT02831153
Title: Effects of Emotional Status on Coronary Flow in Patients Undergoing Coronary Angiography:Multicenter TIMI Frame Count Assessment Study (STRAIN-TIMI Study)
Brief Title: Evaluation of Emotional Status and Coronary Flow Characteristics by TIMI Frame Count Method
Acronym: STRAIN-TIMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ertan YETKIN (Other)
Collaborators: Abant Izzet Baysal University (Other); Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other); Ankara City Hospital Bilkent (Other); Private Yenisehir Hospital (Unknown); Private Gozde Hospital (Unknown); Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, Ertan YETKIN, Director, Clinical Research, Vascular and Molecular Cardiology Society
Organization: Vascular and Molecular Cardiology Society (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Vasmol001
Record Dates: First submitted 2016-07-10; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Ectasia; Slow-Flow Phenomenon; Endothelial Dysfunction; Anxiety; Depression
MeSH Terms: conditions — Coronary Artery Disease; Coronary Aneurysm; No-Reflow Phenomenon; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- normal coronary anatomy (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- coronary artery ectasia (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- slow coronary flow (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- nonobstructive coronary artery disease (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography
- obstructive coronary artery disease (Active Comparator): coronary angiography will be performed by transfemoral or transradial route.
  Interventions: Procedure: coronary angiography

INTERVENTIONS:
Procedure: coronary angiography — Coronary angiography will be performed by transfemoral or transradial approach in all patients. In order to evaluate each coronary artery, at least four views from the left and two views from the right system will be taken.

SUMMARY:
This study evaluates the effects of emotional status on coronary flow in patients undergoing elective coronary angiography. Patients whom undergoing elective coronary angiography will fulfill the Beck Anxiety Inventory, Beck Depression Inventory, State-Trait Anxiety Inventory, Hospital Anxiety and Depression Scale. State Anxiety Inventory will be fulfilled both before the intervention and after 1 hour the patients learned the results of the coronary angiography. The other scales will be performed after 1 hour the patients learned their results. Coronary flow will be assessed by TIMI (Thrombolysis In Myocardial Infarction) frame count method.

ELIGIBILITY:
Inclusion Criteria:

* Patients whom planned elective coronary angiography and accept to be included in the study as a participant

Exclusion Criteria:

* < 18 years, history of prior coronary angiography, history of coronary artery revascularization, acute coronary syndrome patients, atrial fibrillation, heart failure, known systemic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
TIMI frame count method analysis | 1 day

CONTACTS AND LOCATIONS:
Locations (6):
- Turkey (Türkiye) (6):
  - Gulhane Military Medical Academy, Ankara, Kecioren
  - Ankara Numune Training and Research Hospital, Ankara
  - Ankara Research and Training Hospital, Ankara
  - Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Private Gözde Hospital, Malatya
  - Private Yenisehir Hospital, Mersin

IPD SHARING:
Plan to Share IPD: Yes
The results will be made available within 6 months of study completion

REFERENCES:
- [Background] Ozturk S, Yalvac HD, Sivri N, Ozturk HM, Kilic Y, Bulut E, Celik A, Barlas Y, Tengiz I, Yetkin E. Anxiety and depression scores in patients with coronary artery disease and coronary artery ectasia. Int J Cardiol. 2015;186:299-301. doi: 10.1016/j.ijcard.2015.03.305. Epub 2015 Mar 20. No abstract available. PMID 25828141
- [Background] Yalvac D, Ozturk S, Sivri N, Kilic Y, Bulut E, Celik A, Barlas Y, Tengiz I, Yetkin E. Effects of patients anxiety and depression scores on coronary flow in patients with normal coronary arteries. Int J Cardiol. 2015 Feb 1;180:55-7. doi: 10.1016/j.ijcard.2014.11.153. Epub 2014 Nov 26. No abstract available. PMID 25438211
- [Background] Yetkin E, Waltenberger J. Novel insights into an old controversy: is coronary artery ectasia a variant of coronary atherosclerosis? Clin Res Cardiol. 2007 Jun;96(6):331-9. doi: 10.1007/s00392-007-0521-0. Epub 2007 Apr 26. PMID 17453130